CLINICAL TRIAL: NCT02230163
Title: Prevention of Chikungunya Infection in Neonates: Clinical Evaluation of Anti-CHIKV Hyperimmune Intravenous Immunoglobulins
Brief Title: Clinical Evaluation of Anti-CHIKV Hyperimmune Intravenous Immunoglobulins
Acronym: CHIKIVIG-01
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de la Guadeloupe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RBM-PAP-2014/39; 2014-001853-18 (EudraCT Number)
Record Dates: First submitted 2014-08-28; First posted 2014-09-03 (Estimated); Last update posted 2014-11-03 (Estimated); Status verified 2014-08

CONDITIONS: Chikungunya Virus Infection
Keywords: Chikungunya virus; Human anti-CHIKV hyperimmune intravenous immunoglobulins; Neonates
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Biological: anti-CHIKV hyperimmune immunoglobulins — Anti-CHIKV immunoglobulins (CHIKVIg) were purified after the Tégéline manufacturing process from a pool of 583 plasma samples from donors in the convalescent phase of CHIKV infections. Anti-CHIKV hyper immune intravenous immunoglobulin (50 mg/ml) is prepared as a powder to be reconstituted. The therapeutic regimen will consist of 2 doses of 0.5 g/kg 12 hours apart.

SUMMARY:
Chikungunya virus (CHIKV) has been detected in humans in the Caribbean area for the first time in November 2013 (St-Martin Island). By February 2014, the virus had spread to several other Caribbean islands as well as French Guyana, South America. During the outbreak of Chikungunya that affected the Reunion island in 2005/2006, it was observed that the neonatal forms of infections acquired by mother to child transmission during childbirth, were not the exception and were critical. Mother-to-child transmission occurs when the mother is viremic at the time of delivery. The mean duration of viremia after the onset of first clinical symptoms is six days. The rate of mother-to-child transmission is 50%. All neonates contaminated during labor and delivery present with a symptomatic disease and the rate of severe forms is about 50%, primarily due to damage of the central nervous system, often leaving permanent damage (seizures, cerebral palsy).Due to the severity of Chikungunya in neonates and the burden of cerebral palsy, it is imperative to identify a safe and effective preventive and/or curative intervention. Human polyvalent immunoglobulins purified from plasma samples obtained from Chikungunya-convalescent donors exhibit a potent neutralizing activity in vitro. They were evaluated for their preventive and curative effects in a neonatal mouse model of CHIKV infection. After administration of a lethal dose of CHIKV, all neonatal mice that had received immunoglobulins survived while all control animals that had received non hyperimmune immunoglobulins died. In humans, specific human immunoglobulins proved to be effective and safe in neonates born to hepatitis B viremic mothers.

Hypothesis : The investigators hypothesize that the administration of anti-CHIKV hyperimmune human intravenous immunoglobulins to neonates exposed to a high risk of severe form of Chikungunya infection is safe enough to justify its evaluation in an open non randomized trial aimed to confirm the safety and preliminary assess the efficacy of this intervention.

DETAILED DESCRIPTION:
The population to be studied will consist of neonates born to mothers presenting with clinical symptoms of Chikungunya within six days before and two days after childbirth. These neonates will therefore be exposed to a high risk of developing a severe form of Chikungunya infection. In most cases the reality of this risk will have been demonstrated by a positive CHIKV RT-PCR on maternal blood sampled before childbirth.

References to literature and data that are relevant to the trial, and that provide background for the trial.

Chikungunya virus has been detected in humans in the Caribbean area for the first time in November 2013 (St-Martin Island). By February 2014, the virus had spread to several other Caribbean islands as well as French Guyana, South America.

During the outbreak of Chikungunya (CHIK) that affected the Reunion Island in 2005/2006, the neonatal forms of infections acquired by mother-to-child transmission (MTCT) during childbirth, were reported in 50% of viremic mothers and associated with high neonate morbidity. MTCT occurred only when the mother was viremic at the time of delivery. The viremic period begins 2 days before the onset of symptoms and lasts for six days following the first symptoms. In infected neonates contaminated during labor, symptoms appeared after a median incubation period of 4 days. All neonate CHIK cases were symptomatic and the rate of severe forms was about 50%; these severe forms were primarily due to damages to the central nervous system, often leaving permanent damage (seizures, cerebral palsy).

Due to the severity of Chikungunya in neonates and the burden of cerebral palsy, it is imperative to identify a safe and effective preventive and/or curative intervention.

We hypothesize that the administration of hyperimmune human intravenous immunoglobulins to neonates exposed to a high risk of severe form of Chikungunya infection is safe enough to justify its evaluation in an open non randomized trial aimed to confirm the safety and preliminary assess the effectiveness of this intervention.

Although the primary objective of the trial is to assess the safety of hyperimmune human intravenous immunoglobulins in neonates, a clear potential individual benefit is expected for participating neonates, namely a decreased risk of development of a severe form of Chikungunya, especially in terms of high-burden central nervous system complications (seizures, cerebral palsy). This is a major issue since the first case of complicated neonatal Chikungunya has already occurred in Martinique in January 2014 (clinical manifestations included fever, pain, skin rash, and encephalopathy in a four-day-old neonate).

If this trial demonstrates safety and is consistent with potential efficacy of anti-CHIKV hyperimmune intravenous immunoglobulins, this would pave the way to the realization of a phase III trial whose main objective would be to confirm the effectiveness of the strategy, including in other situations, particularly in individuals at risk for severe disease such as exposed neonates and adults with underlying conditions.

This would also be a proof-of-concept for such a therapeutic/preventive strategy in other severe emerging infectious diseases such as arboviral diseases or viral hemorrhagic fevers, as long as no specific drug or vaccine is available.

The risk of developing a severe form in Chikungunya is high in neonates born to CHIKV-viremic mothers. Central nervous system complications represent the most important concern because they are both frequent and frequently associated with permanent brain damages.

To date, no effective therapeutic strategy has been identified in this situation.

The administration of hyperimmune anti-CHICKV intravenous immunoglobulins has proven effective in preventing the development of Chikungunya in a neonatal mouse model.

Several randomized clinical trials demonstrated that intravenous immunoglobulins where safe when administered to neonates and infants.

The first cases of neonatal Chikungunya infection have been identified in French West Indies since the onset of the current outbreak and at least one case was associated with CNS complications.

Pediatricians and neonatologists working in the four hospitals that will participate in the clinical trial have been contacted. They expressed that they are keen to provide a potentially effective therapy to newborns exposed to a high risk of developing of Chikungunya infection and they are convinced that such a treatment would be harmless to neonates, based on their own experience with the use of polyvalent intravenous immunoglobulins.

No specific treatment has been identified to date for Chikungunya infection, especially for severe neonatal forms. While efficacy and safety of anti-CHIKV hyperimmune immunoglobulins have been demonstrated in neonate mice, to date no such study has been performed in humans. Therefore this study would be first to assess this promising therapeutic intervention.

It is also expected that this study will provide new information on the natural history of Chikungunya infection in neonates as well as on the pathophysiology of viral transmission (transplacentally during labor or/and during fetal progression into the genital tract). Actually comparison of quantitative CHIKV RT PCR titers in mother's urine at delivery, placenta, and neonate's blood and other fluids, as well as determination of placental microperfusion markers (placental alkaline phosphatase on cord blood) should shed light on this issue.

Primary endpoint: The primary endpoint will be evaluated in all enrolled neonates. Tolerability and safety of anti-CHIK IVIG will be assessed by evaluating the frequency of patent ductus arteriosus, necrotizing enterocolitis, pulmonary hemorrhage, tachycardia or hypotension during anti-CHIKV IVIG infusion, hemolytic anemia, hyponatremia and ascites.

Secondary endpoints: Secondary endpoints will be evaluated only in neonates born to mothers who had a definite CHIKV-infection.

Primary objective:

The primary objective of the trial is to evaluate the tolerability and safety of anti-CHIKV hyperimmune immunoglobulins given intravenously to neonates exposed to a high risk of MTCT of CHIKV, i.e. born to a mother with definite or possible CHIKV infection at the time of delivery.

Secondary objectives:

The secondary objective of the trial is to evaluate the efficacy of anti-CHIKV hyperimmune immunoglobulins given intravenously in the subgroup of neonates born to mothers with definite CHIKV infection.

Neonates will be classified in one of the following 3 categories:

* Neonatal CHIKV clinical disease:

  * Clinical symptoms consistent with acute CHIKV infection
  * Demonstration of infection based on CHIKV IgM seroconversion and/or identification of CHIKV viremia (positive CHIKV qRT-PCR at Day 3),
* Neonatal CHIKV asymptomatic infection:

  * Absence of any symptom consistent with CHIV infection
  * Demonstration of infection based on CHIKV IgM seroconversion and/or identification of CHIKV viremia (positive CHIKV qRT-PCR at Day 3),
* Neonatal CHIKV infection excluded:

  * Absence of CHIKV IgM seroconversion

Social and Behavioral Science Survey:

In parallel, we will conduct a Social and Behavioral Science survey aimed to assess the factors associated with the parental decision to participate or not in the clinical trial, given its peculiar context (emerging disease, therapeutic intervention in a neonate, invitation to participate in the peri-partum period, short period of time for decision-making.

ELIGIBILITY:
Inclusion Criteria:

* 1. Inclusion criteria in mothers:

  * Clinical symptoms consistent with CHIKV infection (acute-onset high-grade fever combined with bilateral polyarthralgia and no other cause than Chikungunya) during the pre-partum period or within the 48 hours post-partum,
  * Written informed consent obtained,
  * Negative Dengue fever rapid diagnostic test,
  * Blood sampled for CHIKV RT-PCR, processed in emergency, to be used to define 3 diagnosis categories at neonate's birth:
  * positive: definite maternal CHIKV infection,
  * pending: probable maternal CHIKV infection,
  * negative: maternal CHIKV infection excluded.
* 2. Inclusion criteria in neonates:

  * Neonate born to a mother fulfilling ALL maternal inclusion criteria and NO maternal exclusion criteria,
  * Written informed consent signed by both neonate's parents (or legal guardians).

Exclusion Criteria:

* 1. Exclusion criteria in mothers:

  * Delivery more than 6 days after the onset of first symptoms of CHIKV infection,
  * Maternal CHIKV infection excluded,
  * Chronic active HBV infection (positive HBs Ag),
  * HIV infection.
* 2. Exclusion criteria in neonates:

  * Preterm neonate below 28 weeks of gestational age.

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2015-10 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Safety | 30 days
  The primary endpoint will measure tolerability and safety of anti-CHIKV hyperimmune IVIG. It will be evaluated in all enrolled neonates and will be based on the occurrence of the following events:
  * patent ductus arteriosus,
  * ulceronecrotizing enterocolitis,
  * pulmonary hemorrhage,
  * tachycardia, hypotension, decreased O2 saturation during anti-CHIKV IVIG infusion,
  * hemolytic anemia,
  * fluid overload, as indicated by hyponatremia and/or ascites.

SECONDARY OUTCOMES:
Efficacy | 30 days
  The following secondary endpoints will be evaluated only in neonates born to mothers who had a definite CHIKV-infection.
  Neonates will be classified in one of the following 3 categories:
  * Neonatal CHIKV clinical disease:
    * Clinical symptoms consistent with acute CHIKV infection
    * Demonstration of infection based on CHIKV IgM seroconversion and/or identification of CHIKV viremia (positive CHIKV qRT-PCR at Day 3),
  * Neonatal CHIKV asymptomatic infection:
    * Absence of any symptom consistent with CHIV infection
    * Demonstration of infection based on CHIKV IgM seroconversion and/or identification of CHIKV viremia (positive CHIKV qRT-PCR at Day 3),
  * Neonatal CHIKV infection excluded:
    * Absence of CHIKV IgM seroconversion.
  Below is an indicative list of symptoms that are consistent with Chikungunya infection in neonates:
  * Skin rash, severe desquamative disorder, bullous dermatitis,
  * Acral edema
  * Symptoms of encephalopathy/encephalitis : stupor, seizures, impaired sucking

CONTACTS AND LOCATIONS:
Overall Officials: Bruno HOEN, Professor, Principal Investigator — Centre Hospitalier Universitaire de Pointe-à-Pitre
Locations (3):
- France (3):
  - Centre Hospitalier de la Basse-Terre, Basse-Terre, Guadeloupe
  - Centre Hospitalier de Cayenne "Andrée ROSEMON", Cayenne, Guyane
  - CHU de Martinique, Fort-de-France, Martinique